CLINICAL TRIAL: NCT01382342
Title: The Effect of Rasagiline on Cognition in Parkinson's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Principal Investigator, Laura L. Frakey, Clinical Neuropsychologist, Brown University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TNSAZL0016
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; cognition; executive function; rasagiline
MeSH Terms: conditions — Parkinson Disease | interventions — rasagiline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- rasagiline (Experimental): Participants in this arm will receive 1 mg of rasagiline daily for the six month duration of the study.
  Interventions: Drug: Rasagiline
- Placebo (Placebo Comparator): Participants in this group will receive 1 mg of placebo daily for the six month duration of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rasagiline — 1 mg daily
  Other Names: Azilect
  Arms: rasagiline
Drug: Placebo — 1 mg daily
  Arms: Placebo

SUMMARY:
While Parkinson's disease has historically been defined in terms of its motor symptomatology, studies have shown that non-motor deficits form an important part of the syndrome. Cognitive deficits can occur even in the early stages of Parkinson's disease. These deficits are often subtle and do not rise to the level of impairment necessary for a diagnosis of dementia; however these deficits are discernable with neuropsychological testing and may produce subjective complaints of cognitive decline and mild functional difficulties in some patients. The traditional pharmacological interventions for Parkinson's disease have focused on controlling and alleviating motor symptoms with levodopa and dopamine agonists. However, these medications treat the symptoms of PD, but do not alter the course or progression of the underlying disorder. In contrast, rasagiline, an MAO-B inhibitor, has recently shown benefits consistent with a possible disease-modifying effect. Given the positive and intriguing findings seen with treatment with rasagiline, the investigators propose to study the effects of this medication on cognition in patients with mild to moderate stage Parkinson's disease.

Hypotheses:

1. Rasagiline will improve cognitive function, as measured by performance on neuropsychological tests in PD patients who do not suffer from dementia.
2. Rasagiline will not negatively affect neuropsychiatric functioning.

DETAILED DESCRIPTION:
The results of our study found that while participants receiving rasagiline showed some improvements in their motor symptoms, as measured by the UPDRS, no significant changes were found on any of the neuropsychological measures after six months of treatment with rasagiline. Further, the participant group who received placebo also did not show significant change on any of the neuropsychological measures over the six month course of our study. Finally, the cognitive performance of our treatment and placebo groups did not differ significantly from one another at baseline or after six months of study participation.

ELIGIBILITY:
Inclusion Criteria:

* age 40 or older
* able to speak and read English, at least 6 years of formal education
* a diagnosis of PD
* have a family member or caregiver willing to fill out study questionnaires
* Participants will have been on stable medication regimens (no new PD medications and no changes to existing PD medication dosages) for the 4 weeks prior to study enrollment.
* If participants are already taking other Parkinson's medications at time of study enrollment, the dosages of these medications must remain stable throughout study participation.
* Changes to existing Parkinson's disease medications dosages or addition of other medications to treat Parkinson's disease after study enrollment will result in removal from study.
* Participants are allowed to begin non-PD medications or to have changes to their existing non-PD medications if these additions and changes are deemed medically necessary.

Exclusion Criteria:

* currently taking any MAO inhibitor
* currently taking a cognition-enhancing medication such as a cholinesterase inhibitor medication or memantine
* dementia (Mini-Mental Status Exam score below 21/30), significant depression (Beck Depression Inventory- Short Form score >7)
* presence of a another neurodegenerative disorder besides PD
* unstable cardiac disorder, clinically significant hepatic
* lung or renal disease
* In addition, changes to dosages of PD-related medications or the addition of other PD medications during the 6 month study enrollment will result in dismissal from the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Rey Auditory Verbal Learning Test | Change in score from day 1 of study enrollment and score after 6 months of treatment
  This is a 15 item supraspan verbal memory test. This measure assesses immediate memory span, new learning, susceptibility to interference, retention, and recognition memory.

SECONDARY OUTCOMES:
Controlled Oral Word Association Test | day 1 of study enrollment and after 6 months of treatment
  This test evaluates the spontaneous production of words beginning with a given letter of the alphabet under timed conditions. It is used to assess executive functioning.
Animal Fluency | day 1 of study enrollment and after 6 months of treatment
  Participants are asked to produce as many animal names as they can in one minute. This measure assesses executive functioning.
Judgement of Line Orientation from the Repeat Battery for the Assessment of Neuropsychological Status | day 1 of study enrollment and after 6 months of treatment
  This measure assesses spatial perception and orientation without requiring a motor output.
Digit Span from the Wechsler Adult Intelligence Scale- Fourth Edition | day 1 of study enrollment and after 6 months of treatment
  This is a measure of attention and working memory which requires participants to repeat a series of digits forward, in reverse, and to sequence a series of digits.
Trail Making Test | day 1 of study enrollment and after 6 months of treatment
  These are tests of speed for attention, sequencing, mental flexibility, and visual search.
Digit Symbol Modalities Test | day 1 of study enrollment and after 6 months of treatment
  This test assesses cognitive processing speed, and visuomotor coordination and is one of the most sensitive measures of cognitive dysfunction available.
Parkinson's Disease Quality of Life Questionnaire | day 1 of study enrollment and after 6 months of treatment
  The 39-item Parkinson's disease questionnaire (PDQ-39) is one of the most often used instruments to measure treat¬ment effect on quality of life in PD.

CONTACTS AND LOCATIONS:
Overall Officials: Laura L. Frakey, Ph.D., Principal Investigator — Brown University; Joseph Friedman, MD, Principal Investigator — Brown University
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States